CLINICAL TRIAL: NCT06172036
Title: A Multicenter, Multi-cohort, Randomized, Phase II Study of Irinotecan Liposome Combined With 5-FU / LV and Oxaliplatin for Resectable Pancreatic Cancer With or Without Addebelizumab
Brief Title: Irinotecan Liposome for Resectable Pancreatic Cancer With or Without Addebelizumab
Acronym: CAPT-02
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, The chairman of the First Affiliated Hospital of Zhejiang University School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPT-02
Record Dates: First submitted 2023-12-05; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Neoadjuvant Chemotherapy; Resectable Pancreatic Cancer
Keywords: resectable pancreatic cancer; irinotecan liposomes; Adebellizumab
MeSH Terms: interventions — irinotecan sucrosofate; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Preoperative adliberlizumab + irinotecan liposome + oxaliplatin + 5-FU / LV (28 days as one cycle, 2 treatment cycles). Surgery was performed within 2 to 4 weeks after completion of neoadjuvant therapy and addebelizumab + irinotecan liposomes + oxaliplatin + 5-FU / LV (28 days as one cycle, 4 treatment cycles) within 4 to 6 weeks after surgery, followed by maintenance therapy with addebelizumab until disease progression or intolerable toxicity. The cumulative postoperative duration of adbelizumab should not exceed 1 year. Tumor recurrence, safety and survival follow-up was evaluated after completion of the drug.
  Interventions: Drug: irinotecan liposome + oxaliplatin + 5-FU / LV; Drug: Adebellizumab
- Arm B (Experimental): Irinotecan liposome + oxaliplatin + 5-FU / LV (28 days one cycle, 2 treatment cycles), 2-4 weeks after completion of neoadjuvant therapy and 4-6 weeks after surgery, adjuvant irinotecan liposome + oxaliplatin + 5-FU / LV (28 days one cycle, 4 treatment cycles). Tumor recurrence, safety and survival follow-up were performed after the end of the adjuvant treatment phase.
  Interventions: Drug: irinotecan liposome + oxaliplatin + 5-FU / LV
- Arm C (Active Comparator): Upfront surgery, and postoperative adjuvant regimen as with ArmB. Tumor recurrence, safety and survival follow-up were performed after the end of the adjuvant treatment phase.
  Interventions: Drug: irinotecan liposome + oxaliplatin + 5-FU / LV

INTERVENTIONS:
Drug: irinotecan liposome + oxaliplatin + 5-FU / LV — Efficacy and safety of irinotecan liposome combined with oxaliplatin, 5-fluorouracil (5-FU) / leucovorin calcium (LV) with or without adbellizumab for resectable pancreatic cancer
Drug: Adebellizumab — Efficacy and safety of irinotecan liposome combined with oxaliplatin, 5-fluorouracil (5-FU) / leucovorin calcium (LV) with or without adbellizumab for resectable pancreatic cancer
  Arms: Arm A

SUMMARY:
To evaluate the efficacy and safety of irinotecan liposomes with oxaliplatin, 5-fluorouracil (5-FU) / leucovorin (LV) with or without adelizumab for resectable pancreatic cancer by assessing the 12-month EFS rate

DETAILED DESCRIPTION:
For patients with surgically resectable pancreatic cancer who have not received any anti-tumor therapy. To evaluate the efficacy and safety of irinotecan liposomes with oxaliplatin, 5-fluorouracil (5-FU) / leucovorin (LV) with or without adelizumab for resectable pancreatic cancer by assessing the 12-month EFS rate.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years old, male or female;
2. According to the NCCN clinical practice guidelines (2023.V2 version), multidisciplinary and imaging evaluation for patients with resectable pancreatic cancer, resectable defined as: by imaging examination, the criteria of radical resection of tumor is no distant metastasis, the artery (trunk celiac, superior mesenteric artery or common hepatic artery), and the tumor did not invade the superior mesenteric vein and portal vein, or invasion but not more than 180 and the venous contour is normal.
3. Have not received any anti-tumor therapy (including radiotherapy, ablation, chemotherapy, targeted therapy, immunotherapy, etc.) or research drug therapy; 4. At least one measurable lesion must be used as the target lesion (according to the RECIST v1.1 criteria);

5. ECOG：0～1； 6. Expected survival period of 3 months; 7. Main organ function, meeting the following criteria (without receiving any blood components, cell growth factors within the 14 days prior to randomization):

1. Neutrophils 1.5 * 109 / L; platelets 80 * 109 / L; 9 g/dl hemoglobin and 3 g/dl serum albumin;
2. The upper limit of total bilirubin is 1.5 times (biliary obstruction allows biliary drainage); the upper limit of ALT and AST is 3 times (for patients of liver metastasis, it can be relaxed to 5 times the upper limit of normal);
3. The upper limit of normal serum creatinine is 1.5 times, and the creatinine clearance is 60ml / min;
4. The upper limit of INR is 1.5 times and the upper limit of APTT is 1.5 times (for stable doses of anticoagulant therapy such as low molecular weight heparin or warfarin and INR can be screened within the expected treatment range of anticoagulant);
5. ECG: QTcF 450ms (male), 470ms (female);
6. Cardiac color ultrasound: LVEF (left ventricular ejection fraction) 50%; 8. Women of childbearing age must have a negative blood pregnancy test within 3 days before randomization and be willing to use appropriate contraception during the trial and within 6 months of treatment. For men, it should be surgical sterilization, or consent to use appropriate methods of contraception during the study period and within 3 months after the end of treatment; 9. Subjects volunteered to join the study and signed the informed consent form.

Exclusion Criteria:

1. Patients with pancreatic cancer arising from non-pancreatic ductal epithelium, including pancreatic neuroendocrine carcinoma, pancreatic acinar cell carcinoma, pancreatic pancreoblastoma, and solid-pseudopapillary tumors;
2. Patients with known central nervous system metastases;
3. Severe gastrointestinal dysfunction (bleeding, obstruction; inflammation greater than grade 2; diarrhea greater than grade 1);
4. Within 2 weeks before randomization, the third space effusion (such as a large amount of pleural fluid) (no intervention after removing the drainage tube);
5. Patients with clinical symptoms of ascites, requiring puncture, drainage, who have received ascites drainage within the previous 3 months (only a small amount of ascites on imaging and controllable, except those without clinical symptoms);
6. Current subjects with interstitial pneumonia or interstitial lung disease, or a history requiring hormonal therapy, or other pulmonary fibrosis, mechanical pneumonia (e. g., bronchiolitis obliterans), pneumoconiosis, drug-related pneumonia, idiopathic pneumonia, idiopathic pneumonia or active CT during screening that may interfere with the judgment and management of immune-related pulmonary toxicity; active tuberculosis;
7. Patients with active autoimmune disease or a history of autoimmune disease that may relapse [including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, optis, enteritis, vasculitis, nephritis, hyperthyroidism, reduced thyroid function (only controlled by hormone replacement therapy can be enrolled)]; skin diseases without systemic treatment, such as vitiligo, psoriasis, alopecia, controlled type I diabetes or asthma in childhood has been completely alleviated in adults without any intervention;
8. Known peripheral neuropathy (CTCAE Grade 3);
9. Known dihydropyrimidine dehydrogenase (low activity) or deficiency;
10. Severe infection (CTCAE> 2), such as severe pneumonia, bacteremia, infectious complications, requiring hospitalization, occurred within 4 weeks of randomization; symptoms and signs of infection within 2 weeks of randomization (except in cases of prophylactic antibiotics);
11. Received any of the following treatments:

(1)Concomitant medication containing CYP3A4, CYP2C8 strong inhibitor / strong inducer or strong UGT1A1 inhibitor within 2 weeks before randomization; (2)Immunosuppressants or systemic hormone therapy within 2 weeks prior to randomization to achieve immunosuppressive purposes (dose> 10mg prednisone / day or other efficacy hormones); (3)Received radiation therapy within 2 weeks before randomization; (4)Receiving major surgery (such as thoracotomy, laparotomy, etc.) within 4 weeks before randomization; (5)Have received any other clinical study drug treatment within 4 weeks before randomization, except for an observational (non-interventional) clinical study or interventional clinical study follow-up.

12. Abnormal coagulation, bleeding tendency or undergoing thrombolytic or anticoagulant therapy. Prophylactic use of low-dose aspirin (100mg / day), low molecular weight heparin (enoxaparin 40mg / day and other low molecular weight heparin at its equivalent doses) is allowed; 13. cardiac clinical symptoms or diseases that are not well controlled, such as: (1) heart failure; (2) unstable angina; (3) myocardial infarction within 6 months; (4) patients with clinically significant supraventricular or ventricular arrhythmias who need treatment or intervention; 14. Malignant tumors other than pancreatic cancer within 5 years before randomization, except for adequately treated cervical carcinoma in situ, skin basal cell, or squamous epithelial cell carcinoma; 15. Those known to be allergic to PD-L1, irinotecan liposomal, other liposomal products, oxaliplatin, 5-FU, leucovorin and any of the components of the above products; 16. Those known to have acquired immune deficiency syndrome (AIDS) or HIV test positive, active syphilis; 17. A clear past history of neurological or psychiatric disorders, including epilepsy or dementia; 18. By the judgment of the investigator, the subject has other factors that may be forced to terminate the study, such as non-compliance protocol, with other serious diseases (including mental illness) need to combine treatment, clinical significant laboratory value seriously abnormal, family or social factors, may affect the safety or trial data collection of subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
12-month EFS rate | Up to 2 years.
  the proportion of subjects with EFS events within one year.

SECONDARY OUTCOMES:
Overall Survival | Up to 2 years.
  Defined as the time from random to death from any cause
Event free survival | Up to 2 years.
  Defined as the time from randomization to disease progression, disease recurrence or death from any cause.
Disease free survival | Up to 2 years.
  Defined as the time from randomization to disease recurrence or death from any cause.
Objective response rate | Up to 2 years.
  Evaluation of the ORR by the investigator per RECIST v1.1 criteria means the proportion of subjects with the best overall efficacy of CR or PR. If the efficacy reaches CR and PR, the subject must be reviewed 4 weeks after the initial evaluation.
R0 resection rate | Up to 2 years.
  Defined as the proportion of subjects assessed as R0 resection.
Incidence of Treatment-Emergent Adverse Events | Up to 2 years.
  Incidence of Adverse events (AEs) / serious adverse events (SAEs) (as per NCI-CTCAE 5.0)

IPD SHARING:
Plan to Share IPD: No